CLINICAL TRIAL: NCT03529240
Title: Kinesiology Taping in Duchenne Muscular Dystrophy: Effects on Performance, Gait Characteristics, and Energy Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güllü AYDIN, Research Assistant Güllü AYDIN, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KA-17070
Record Dates: First submitted 2018-05-06; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Performance; Energy; Gait; Duchenne Muscular Dystrophy
Keywords: kinesiology taping; performance; energy consumption; gait; Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kinesiology taping (Experimental): After performing the baseline assessments, kinesiology taping with facilitation technique was applied on bilateral quadriceps and tibialis anterior muscles of children. In both applications, the first and last 5 cm section of the bands were used as anchor and no tension was applied.
  Interventions: Device: Kinesiology Taping

INTERVENTIONS:
Device: Kinesiology Taping — Kinesiology taping (KT) which was developed by Dr. Kenzo Kase, is a new application of elastic and adhesive taping. KT is applied by specialized physiotherapists and physicians. This type of taping is a very frequently used technique to accelerate recovery after musculoskeletal injuries. Also, this technique is usually used as an alternative to athletic taping to support fascias, muscles, and joints for many purpose such as positioning, inhibition, and fascilitation

SUMMARY:
Investigators investigated that the effects of kinesilogy taping on performance, energy consumption and gait characteristics in patients with Duchenne Muscular Dystrophy

DETAILED DESCRIPTION:
Forty-five patients from Level 1 and 2 according to the Brooke Lower Extremity Functional Classification were included in the study. Performance was assessed by measuring the distance in 6-minute walk test (6MWT) and the duration of timed performance tests; energy consumption by Physiological Consumption Index (PCI), and gait characteristics by footprint method on powdered ground at baseline. Kinesiology taping with facilitation technique was applied on bilateral quadriceps and tibialis anterior muscles and the assessments were repeated 1 hour after application. The comparison between before and after taping was analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Duchenne Muscular Dystrophy diagnosis,
* age 5 to 14 years,
* able to cooperate with instructions of physiotherapist,
* able to walk independently,
* climb 4 steps independently/with minimal support from handrails.

Exclusion Criteria:

* severe contracture at lower extremities,
* other disease except for DMD, and
* history of any injury or orthopaedic/neurologic surgery within the past 6 months.

Ages: 5 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2017-08-05 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Test | 6 minute
  Six Minute Walk Test was used commonly in DMD were found to be valid, reliable and easy to apply in the clinic. Children were asked to walk during 6 minutes as fast as they can at a corridor specified by two cones and walking distances were recorded as meter (m) for 6MWT. The time passed during timed performance tests were recorded as seconds.

SECONDARY OUTCOMES:
Energy Consumption | 6 minutes
  Physiologic Consumption Index (PCI) was used to evaluate energy consumption of children during 6MWT. energy consumption was calculated by using the formula of PCI (walking heart rate)-(resting heart rate)/(walking speed)
Gait | 2 minutes
  Gait analysis of the children was performed by footprint method on 10-meters powdered floor. First and last 2 meters of this floor were dissociated from the assessment, and both the right and left stride lengths, both right and left foot angles, and stride width were analyzed in the middle 6-meter section.. Stride length was measured by measuring the distance between right and left midpoint heels. Double stride length was sum of right and left stride length. Stride width was measured by horizontal distance between heel midpoints. Foot angles were measured by a goniometer considering the line between the first and second metatarsal heads and the heel midpoints of both feet separately 24. The number of steps during 6MWT was also calculated by pedometer (Omron, Walking style One 2.0 HJ-320-E) and recorded.
Timed Performance Test | 10 minutes
  Ascending-descending standard 4 steps, walking 10m, standing from lying position were used in order to assess the performance of children.The time passed during timed performance tests were recorded as seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Güllü Aydın, R.A, Principal Investigator — Hacettepe University; İpek Alemdaroğlu Gürbüz, Assoc. Prof., Study Director — Hacettepe University; Öznur Yılmaz, Prof., Principal Investigator — Hacettepe University; Ayşe Karaduman, Prof., Principal Investigator — Hacettepe University; Numan Bulut, R.A, Principal Investigator — Hacettepe University; Haluk Topaloğlu, Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)